CLINICAL TRIAL: NCT01091324
Title: The Reno-protective and Cardiovascular Effect of Dextromethorphan and Silymarin in Patients With Chronic Kidney Disease
Brief Title: Dextromethorphan and Silymarin in Chronic Kidney Disease (CKD) Patients
Acronym: CKD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Junne-Ming Sung, National Cheng Kung University Hospital (NCKUH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-97-108
Record Dates: First submitted 2010-02-09; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Proteinuria
Keywords: CKD, proteinuria, dextromethorphan, silymarin; patients with 15 ml<eGFR< 60ml and 0.5 g/day<proteinuria<3g/day
MeSH Terms: conditions — Proteinuria | interventions — Dextromethorphan; Silymarin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dextromethorphan (Active Comparator)
  Interventions: Drug: Dextromethorphan
- Silymarin (Active Comparator)
  Interventions: Drug: Silymarin
- sugar pill (Placebo Comparator)
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Dextromethorphan — 60 mg, bid
  Arms: Dextromethorphan
Drug: Silymarin — 150 mg , tid
  Arms: Silymarin
Drug: sugar pill — placebo
  Arms: sugar pill

SUMMARY:
The investigators test the renal and cardiovascular protective effects dextromethorphan and silymarin on patients with the proteinuric chronic kidney diseases, who enrolled in our clinical trial, had progressing kidney diseases and merit aggressive anti-inflammatory therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Stage 3 or 4 chronic kidney disease as measured by a Modification in Diet in Renal Disease Study (MDRD) estimate of between 15 ml/min and 59 ml/min and and 0.5 g/day<proteinuria<3g/day.
2. Age between 18 and 75 years old.
3. Patients without hospitalization for cardiac or infection related morbidity over the previous 2 months(due to the potential confounding effects on baseline study variables).
4. Patients who are able to provide consent to participate in the study.-

Exclusion Criteria:

1. patients will significant mental illness, pregnant women, and other vulnerable populations.
2. Patients with active hepatic disease and/or ALT > 2.5 times upper limit of normal.
3. Patients with history of congestive heart failure and NYHA Class III-IV symptoms at any time.
4. Patients for whom living donor renal transplantation is already scheduled or in the process of being evaluated, as these patients will be unlikely to complete study protocols before transplantation.
5. Patients with severe co-morbid conditions (eg, symptomatic hepatic cirrhosis, metastatic cancer, HIV infection with AIDS).
6. Patient with active inflammatory process (eg., SLE, rheumatoid arthritis, gout) for which they are currently receiving immune modulating medications.
7. Patients who are on corticosteroid therapy.
8. Patients who do not consent to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
change of eGFR | 4 months
  Use MDRD-simplified equation
Change of Urine TP/Cr | 4 months
Change of serum hsCRP | 4 months
Change of urine TGF-beta/Cr level | 4 months
  fibrotic marker of kidney
Endothelial function | 4 months
  by Flow-mediated dilatation mesured by Crdiovascular ultrasound

SECONDARY OUTCOMES:
Leukocyte ROCK activity | 4 months
  Measure leukocyte Ro kinase activity by western blotting This is an indicator of cardiovascular function
Blood MDA level | 4 months
  Indicator of oxidative stress
Blood TGF-beta | 4 months
  By Elisa
Urine MCP-1/Cr level | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Junne-Ming Sung, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Taian, Taiwan, Taiwan